CLINICAL TRIAL: NCT01839578
Title: Regional Citrate Versus Systemic Heparin Anticoagulation for Super High-flux Continuous Hemodialysis in Septic Shock: Effect on Middle Molecular Weight Molecules Clearances
Brief Title: Citrate Versus Heparin Anticoagulation: Effect on Molecules Clearances
Acronym: RCA-SHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012.724
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Septic Shock
Keywords: cytokines; blood purification; super high flux hemodialysis
MeSH Terms: conditions — Shock, Septic | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RCA Group (Experimental): SHF-CVVHD with regional citrate anticoagulation
  Interventions: Drug: Anticoagulation to prevent clotting of the extracorporeal circuit. (regional citrate anticoagulation)
- Heparin group (Experimental): SHF-CVVHD with systemic heparin anticoagulation
  Interventions: Drug: Anticoagulation to prevent clotting of the extracorporeal circuit (Unfractionated heparin)

INTERVENTIONS:
Drug: Anticoagulation to prevent clotting of the extracorporeal circuit. (regional citrate anticoagulation) — Anticoagulation to prevent clotting of the extracorporeal circuit. Unfractionated heparin and regional citrate anticoagulation will be compared.
  Ci-Ca protocole for MultiFiltrate® CRRT machine :
  * 4% trisodium citrate solution
  * Calcium chloride solution (100 mmol/L)
  * Dialysate flow rate: 35 ml/kg/h
  * Blood flow rate: adjusted to maintain a ratio blood flow rate / dialysate flow rate of 3
  * Citrate infusion titrated to maintain postfilter ionized calcium between 0.25 and 0.35 mmol/L.
  * Calcium chloride infusion titrated to maintain systemic ionized calcium between 1.12 and 1.2 mmol/L.
  * Blood flow adapted to the acid-base status
  Arms: RCA Group
Drug: Anticoagulation to prevent clotting of the extracorporeal circuit (Unfractionated heparin) — Anticoagulation to prevent clotting of the extracorporeal circuit. Unfractionated heparin and regional citrate anticoagulation will be compared.
  * Continuous infusion of unfractionated heparin: starting infusion rate at 600 IU/h then adjusted to maintain partial thromboplastin time at 1-1.4 times the normal value.
  * Standard dialysate for CRRT : Prismasol® K2 solution
  * Dialysate flow rate: 35 ml/kg/h
  * Blood flow rate: adjusted to maintain a ratio blood flow rate / dialysate flow rate of
  Arms: Heparin group

SUMMARY:
Sepsis is responsible for 50% of all acute kidney injury (AKI) in intensive care units (ICUs), contributing greatly to multiple organ dysfunction syndrome (MODS). Special types of continuous renal replacement therapies (CRRT) have been proposed as adjuvant therapies for septic shock due to their ability to remove middle molecular weight molecules such as inflammatory mediators involved in MODS pathophysiology. These therapies are called extracorporeal " blood purification " therapies.

When CRRT is used, an anticoagulation is required to prevent clotting of the extracorporeal circuit, possibly causing bleeding in selected patients. Many anticoagulation strategies have been proposed and the most commonly used in 2013 is still unfractionated heparin. Regional citrate anticoagulation (RCA) is an interesting alternative as it dramatically decreases the bleeding risk.

The investigators hypothesize that the use of citrate with Super High Flux Continuous Veno-Venus Hemodialysis (SHF-CVVHD) would be highly beneficial over time by preserving the filter effectiveness via limiting protein adhesion (which subsequently reduces filter pore sizes (protein cake)), as compared to heparin. Consequently, higher clearances of the inflammatory mediators could be maintained over time with citrate as compared to heparin anticoagulation. In other words, for the same duration of filter use, middle molecular weight molecules and cytokines clearances would be greater with citrate as compared to heparin. To test this hypothesis, the investigators will perform a clinical randomized controlled trial which aim would be to compare middle molecular weight molecules and cytokines clearances in SHF-CVVHD using RCA versus systemic heparin anticoagulation in septic patients with AKI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female critically ill patients over the age of 18 years old
* Acute Kidney Injury requiring CRRT defined using the Risk, Injury, Failure, Loss, End-stage renal disease (RIFLE) classification with criterion I or worse.
* Septic shock as defined by the American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference.
* Written informed consent obtained from the patient or a patient's legal representative
* Patient patient's legal representative able to agree to patient's enrollment in the study with informed consent.

Exclusion Criteria:

* Pregnancy
* Participation in another research study protocol
* Known heparin induced thrombopenia or contraindication to heparin
* Pre-existing chronic renal failure on chronic dialysis
* Therapeutic anticoagulation with heparin for another reason (e.g. chonic arrhythmia)
* Severe liver failure (15% prothrombin time)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-11 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Middle molecular weight molecules clearances | 18 months
  At each time point of the study (T=1h,T=4h,T=12h,T=24h, T=48h, and T=72h), blood and post-filter samplings will be taken in order to calculate kappa and lambda light chains of immunoglobulin clearances.

SECONDARY OUTCOMES:
Clearances of cytokines and molecules of interest | T=1h,T=4h,T=12h,T=24h, T=48h, and T=72h
  At each time point of the study (T=1h,T=4h,T=12h,T=24h, T=48h, and T=72h), sampling will be simultaneously collected from blood and post-filter in order to determine cytokines (IL-1 ra, IL-10, IL-6, IL-8, β2microglobuline), urea, creatinine and albumin clearances.
Hemodynamic parameters | T=1h,T=4h,T=12h,T=24h, T=48h, and T=72h
  At each time point of the study (T=1h,T=4h,T=12h,T=24h, T=48h, and T=72h), clinical data and blood sampling will be collected in order to assess mean arterial pressure, heart rate, vasopressor requirement and lactate level.
Respiratory parameters | (T=1h,T=4h,T=12h,T=24h, T=48h, and T=72h),
  At each time point of the study (T=1h,T=4h,T=12h,T=24h, T=48h, and T=72h), PaO2/FIO2 ratio will be measured by blood sampling and clinical data collection.
mortality | 28th day

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation - Pavillon P, Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078